CLINICAL TRIAL: NCT06615973
Title: Screening for Social Determinants of Health (SDOH) and Cognitive Function in Individuals With History of Stroke
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001861; 001861-N
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05-16

CONDITIONS: Stroke; Brain Disease; Vascular Diseases; Cerebrovascular Disorder
Keywords: Stroke; Social Determinants of Health; Cognition; cerebrovascular health; Magnetic Resonance Imaging (MRI); vascular health
MeSH Terms: conditions — Stroke; Brain Diseases; Vascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Participants who were enrolled in Natural History Study in past 6 years

SUMMARY:
Background:

Stroke is the fifth leading cause of death in the United States. It is also a leading cause of disability. More than 70% of people who survive strokes have mental impairment or dementia. Medical factors, such as the severity of the stroke, affect whether a person will have mental impairment afterward. But social factors, such as education and ethnicity, seem to play a role as well. Researchers want to learn more about how social and lifestyle factors affect a person s chances of maintaining mental functions after a stroke.

Objective:

To better understand how social and lifestyle factors affect the risk of mental impairment after a stroke.

Eligibility:

People aged 18 years and older who had a stroke and a brain scan while they were enrolled in NIH Study 01N0007 (Natural History of Stroke Study).

Design:

Participants will have 1 study visit, by telephone. The call will last about 45 minutes. Participants will talk about their health since their stroke. They will answer questions about themselves. Topics will include:

* Their race
* Education
* Ethnicity
* Employment
* Marital status
* Residence address
* Recent health history
* Medical insurance

They will have tests of their memory, attention, and language skills. They will repeat numbers and words forward and backward.

Researchers will look at the data and imaging scans collected during participant s enrollment in NIH Study 01N0007. This data will include:

* The hospital that first saw the participant at the time of their stroke.
* The type of imaging that was first used then.
* The primary diagnosis at admission.
* Other medical details.

DETAILED DESCRIPTION:
Study Description:

Clinical health outcomes and the likelihood of post stroke cognitive impairment and dementia (PSCID) can greatly vary following stroke incidence. Thus, developing a better understanding of what characteristics might provide resilience and enrich post-stroke recovery is of utmost importance. The NINDS Natural History of Stroke study (01N0007) was designed with the intention to generate natural history data of participants with or at-risk for acute stroke, transient ischemic attack (TIA), and other disturbances of cerebrovascular circulation. Through use of participants enrolled in the Natural History of Stroke study within the past six years, we aim to characterize social determinants of health (SDOH) and present-day cognitive function in this cohort. Following the collection of these data, we will examine how the core volume of acute supratentorial infarcts relates to post-stroke function as measured by the NIHSS, and how this association is modified based upon SDOH features and independent of treatment.

Objectives:

* To characterize SDOH and assess if such characteristics modify the relationship between MRI core infarct volume and post-stroke function (i.e., NIHSS) at baseline and/or discharge. Resilience will thus be assessed by evaluating how specified SDOH modify the correlation between MRI core infarct volume and NIHSS.
* To assess present cognitive function and assess if SDOH modify the relationship between MRI core infarct volume and present-day cognition. Resilience will thus be assessed by evaluating how SDOH modify the correlation between infarct volume and present-day cognition.
* To assess if SDOH modify the relationship between poststroke function (i.e. NIHSS) at baseline and/or discharge with present-day cognition. Resilience will thus be assessed by evaluating how SDOH modify the correlation between NIHSS and present-day cognition.

Endpoints:

The primary purpose of this study is to assess SDOH and cognitive function in participants who have had a stroke in the past six years. To this end, the primary study outcomes will be post-stroke function as defined by NIHSS and present-day cognitive function.

* Primary Endpoint: Association between MRI core infarct volume and post-stroke function (i.e. NIHSS) as modified by SDOH.
* Secondary Endpoints: Association between MRI core infarct volume and present-day cognitive function as modified by SDOH.
* Exploratory Endpoint: Association between post-stroke function (i.e. NIHSS) and present-day cognitive function as modified by SDOH.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Adults aged 18 or older.
* Previous participant in the Natural History of Stroke with an interpretable baseline MRI scan, NIHSS measured at baseline or discharge, and admission diagnosis of ischemic stroke.
* Fluent in English or Spanish

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

* Modified Rankin Scale (mRS) = 6 at any follow-up (usually up to 90 days) in the Natural History of Stroke study (mRS = 6 indicates the participant is dead).
* Is pregnant per self-report

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants that were previously enrolled (and had a MRI) within the past 6 years in the NINDS Stroke Branch Natural History study will be recruited for enrollment in the present study. Estimated to be 450 participants (18 and older). Study will consist of one phone call and during the phone call, population will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Post-stroke function as defined by NIH Stroke Scale (NIHSS) | NIHSS and core infarct volume gathered at time of enrollment in Natural History of Stroke study, SDOH gathered at present
  Will use linear regression models to assess association between core infarct volume and post stroke function (as defined by NIHSS) as modified by SDOH

SECONDARY OUTCOMES:
Present-day cognitive function | SDOH and present-day cognitive function gathered over phone (present "visit"), other data (including core infarct volume) gathered at time of Natural History of Stroke enrollment
  Will use linear regression models to assess association between core infarct volume and present-day cognition as modified by SDOH

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca F Gottesman, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identifiable Individual participant data will be made available across NIMH Data Archive (NDA), an institutional repository supported by NIMH that makes clinical, imaging, and neurosignal data accessible and sharable across scientific domains. NDA provides infrastructure for sharing research data, tools, methods, and analyses enabling collaborative science and discovery. De-identified subjects data, harmonized to a common standard, are available to qualified researchers. Summary data are available to all. De-identifiable data will be made available as soon as possible or at the time of associated publication. The NDA mission is to accelerate scientific research and discovery through data sharing, data harmonization, and the reporting of research results.
Supporting Information: Study Protocol, ICF
Time Frame: De-identifiable data will be made available as soon as possible or at the time of associated publication, whichever comes first.@@@@@@
Access Criteria: Requests for data access will need to adhere to the standard processes per each repository. These repositories allow for querying and access to shared datasets.

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Chalela JA, Kidwell CS, Nentwich LM, Luby M, Butman JA, Demchuk AM, Hill MD, Patronas N, Latour L, Warach S. Magnetic resonance imaging and computed tomography in emergency assessment of patients with suspected acute stroke: a prospective comparison. Lancet. 2007 Jan 27;369(9558):293-8. doi: 10.1016/S0140-6736(07)60151-2. PMID 17258669
- [Background] Clark DG, Boan AD, Sims-Robinson C, Adams RJ, Amella EJ, Benitez A, Lackland DT, Ovbiagele B. Differential Impact of Index Stroke on Dementia Risk in African-Americans Compared to Whites. J Stroke Cerebrovasc Dis. 2018 Oct;27(10):2725-2730. doi: 10.1016/j.jstrokecerebrovasdis.2018.05.048. Epub 2018 Aug 1. PMID 30076114
- [Background] Douiri A, Rudd AG, Wolfe CD. Prevalence of poststroke cognitive impairment: South London Stroke Register 1995-2010. Stroke. 2013 Jan;44(1):138-45. doi: 10.1161/STROKEAHA.112.670844. Epub 2012 Nov 13. PMID 23150656
- [Background] El Husseini N, Katzan IL, Rost NS, Blake ML, Byun E, Pendlebury ST, Aparicio HJ, Marquine MJ, Gottesman RF, Smith EE; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Radiology and Intervention; Council on Hypertension; and Council on Lifestyle and Cardiometabolic Health. Cognitive Impairment After Ischemic and Hemorrhagic Stroke: A Scientific Statement From the American Heart Association/American Stroke Association. Stroke. 2023 Jun;54(6):e272-e291. doi: 10.1161/STR.0000000000000430. Epub 2023 May 1. PMID 37125534
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001861-N.html